CLINICAL TRIAL: NCT07048132
Title: Validity and Reliability of the Turkish Version of the Headache Screening Questionnaire
Brief Title: Turkish Version of the Headache Screening Questionnaire
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Tanyel Saraçoğlu, Medical doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/169
Record Dates: First submitted 2025-06-21; First posted 2025-07-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Tension Type Headache; Headache
Keywords: migraine; tension type headache; headache; headache screening questionare; validation; reliability
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with headache
  Interventions: Diagnostic Test: Headache Screening Questionare

INTERVENTIONS:
Diagnostic Test: Headache Screening Questionare — The Headache Screening Questionnaire (HSQ) is a 10-item tool developed to screen for migraine and tension-type headache (TTH), based on the ICHD-3 beta criteria.
  Each item reflects a diagnostic criterion for migraine or TTH. Participants complete the HSQ and are also evaluated by a neurologist for diagnosis.
  A score of 6 or higher suggests "probable migraine" or "probable TTH."

SUMMARY:
This multi-center, nationwide study aims to evaluate the validity and reliability of the Turkish version of the Headache Screening Questionnaire (HSQ-TR). The 10-item questionnaire is designed to screen for migraine and tension-type headache in individuals with headache complaints.

Participants presenting with headache will be enrolled. Each participant will first complete the HSQ-TR and then be examined by a neurologist who will provide a diagnosis according to the ICHD-3 beta criteria. The questionnaire results will be compared with the neurologist's diagnoses to assess criterion validity, including sensitivity, specificity, and agreement.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over who present with headache complaints (migraine or tension-type) and voluntarily agree to participate

Exclusion Criteria:

* Individuals with severe psychiatric disorders, illiteracy in Turkish, or significant cognitive impairment preventing comprehension of the scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) presenting with headache complaints (migraine or tension-type headache) at outpatient neurology clinics in participating hospitals. Participants must be literate in Turkish and cognitively capable of completing self-report questionnaires. A total of 100 patients will be enrolled across multiple centers in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
ICHD-3 Beta Classification | Day 1, Two weeks later control
Headache Screening Questionare | Day 1,Two weeks later control

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Gürsoy, Medical Doctor, Principal Investigator — Ümraniye Research and Training Hospital

IPD SHARING:
Plan to Share IPD: No